CLINICAL TRIAL: NCT04688099
Title: A Single-center Observational Study of the Relationship Between Sleep, Synovial Fluid Cytokine Profiles, & Outcomes of ACL Reconstruction
Brief Title: Synovial Fluid Sleep Study
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-01872
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study of the relationship between perioperative sleep time/quality, synovial fluid cytokine profiles, and clinical outcomes of primary ACL reconstruction with BPTB autograft in 50 subjects. Sleep during the week before and month after surgery will be assessed using Fitbit smartwatch and sleep diary. Synovial fluid sampled preoperatively, intraoperatively, and postoperatively will be analyzed for levels of pro- and anti-inflammatory cytokines. Postoperative knee pain and function will be assessed until 2 years post-op using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Undergoing primary ACL reconstruction with BPTB autograft for acute ACL tear, with or without concomitant meniscectomy
3. Presenting within 2 weeks of injury and undergoing reconstruction within 8 weeks of injury

Exclusion Criteria:

1. History of blood-borne diseases including HIV, HBV, HCV, HTLV, or syphilis
2. Pregnant
3. Multiligamentous knee injury
4. Concomitant meniscal repair, meniscal allograft transplantation, osteotomy, or repair of focal chondral defect (e.g., osteochondral autograft transfer system, osteochondral allograft, matrix-induced autologous chondrocyte implantation)
5. Prior ipsilateral knee surgeries or injuries
6. Primary sleep disorders including insomnia, sleep apnea, or restless legs syndrome
7. Uncontrolled psychiatric disorders with sleep disturbance
8. Night shift work
9. Travel with time zone change within three weeks of surgery
10. Systemic inflammatory disease
11. Autoimmune disease
12. Immunomodulatory drug use
13. Chemotherapy within a year before surgery
14. Intra-articular injection within 3 months before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adults with acute ACL tear undergoing primary reconstruction with BPTB autograft
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Year 2
  KOOS is a survey is meant to track how the participant feels about their knee and how well they are able to perform their usual activities. There are six categories in the survey: Symptoms, Stiffness, Pain, Function/Daily Living, Function/Sports, Quality of Life.
  1. Symptoms category consists of 5 questions, ranked from "never" to "always" (0-5).
  2. Stiffness category consists of 2 questions, ranked from "none" to "extreme" (0-5).
  3. Pain category consists of 9 questions, ranked from "none" to "extreme" (0-5).
  4. Function/Daily Living category consists of 17 questions, ranked from "none" to "extreme" (0-5).
  5. Function/Sports category consists of 5 questions, ranked from "none" to "extreme" (0-5).
  6. Quality of Life category consists of 4 questions, ranked from "not at all" to "extremely, constantly, totally" (0-5).
  The total range of score is 0-210. The lower the score, the better they feel about their knee and performance of usual activities.

SECONDARY OUTCOMES:
Score on Lysholm Knee Scoring Scale | Year 2
  The Lysholm Knee Scoring Scale consists of 35 common complaints which people frequently have with their knee problems. Participants will check each statement which best describes their condition -- each statement is assigned a particular score, and those scores are added together to obtain the total score out of 100 (total range: 0-100). A higher score indicates more knee problems.
VAS Score for Anterior Knee Pain | Year 2
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The total score range is 0-10; the higher the score, the worse the pain.
Knee Range of Motion | Year 1
  Knee range of motion (maximal flexion and extension) will be measured bilaterally using a goniometer.
Thigh Circumference | Year 1
  Thigh circumference will be measured bilaterally.
Concentration of Synovial Fluid Cytokines | Year 1
  Synovial fluid from the injured knee will be sampled preoperatively, intraoperatively, and postoperatively and analyzed for levels of the following pro- and anti-inflammatory cytokines using multiplex magnetic bead immunoassay or ELISA: matrix metalloproteinase (MMP) 3, tissue inhibitor of metalloproteinase (TIMP) 1, TIMP-2, interleukin-1 receptor antagonist (IL-1ra), IL-6, monocyte chemotactic protein (MCP) 1, macrophage inflammatory protein (MIP) 1beta/CCL4, RANTES (regulated upon activation, normal T cell expressed and secreted), vascular endothelial growth factor (VEGF), and basic fibroblast growth factor (bFGF/FGF-2).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to eric.strauss@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.